CLINICAL TRIAL: NCT03418103
Title: System to Avoid Fall Events: A Descriptive Comparison Study Evaluating the Quantitative Impact of Using Thermal Imaging to Monitor At-risk Patients.
Brief Title: System to Avoid Fall Events
Acronym: SAFE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rinicare Ltd (Industry)
Collaborators: University Hospitals of Morecambe Bay NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 999
Record Dates: First submitted 2018-01-25; First posted 2018-02-01 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-01

CONDITIONS: Accidental Fall

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Thermal imaging analysis of participant position in a hospital bed — The SAFE sensor system will use thermal imaging to detect and identify a participant's position relative to the edges of the hospital bed. If a dangerous position is identified, an alarm notification will be sent to the ward staff to allow them to take pre-emptive action to prevent the participant's situation from evolving into a fall event.

SUMMARY:
Rinicare Ltd, a Lancaster-based SME, and University Hospitals of Morecambe Bay Trust (UHMB) will collaborate on a research study to determine the feasibility, suitability, and acceptability of the Rinicare developed SAFE (System to Avoid Fall Events) fall prevention and detection system in a hospital environment. The study is designed to determine if the implementation of the SAFE system will help clinicians to prevent in-patient falls from hospital beds. In-patient falls are a serious problem with more than 245,000 incidents reports in 2015-2016. 77% of these falls involve a patient over the age of 65, and the injuries patients suffer due to falls is estimated by NICE to cost the NHS £2.3B annually. This study will test the performance of the SAFE technologies against the current interventions to prevent falls, and it will investigate the impact of the SAFE technology on the workflow of the carers.

The SAFE study is designed as a comparison study combining a descriptive, quantitative methodology measuring the number of fall events with a normative analysis of the qualitative aspects experienced by the clinicians using the SAFE system during the project period.

The primary research objective of this study is to determine if the implementation of the SAFE system will quantifiably reduce the number of fall events in the ward compared to a similar control period. The secondary research objective is to determine if the SAFE system has a positive or a negative impact on the ward staff's workflow, i.e. the ability of the ward staff to provide care to the patients.

ELIGIBILITY:
Inclusion Criteria:

Patients who are deemed by the ward clinicians to be at risk of falling from the bed due to one or more of the following reasons:

* Frailty due to old age (E.g. 65 years or older)
* Frailty due to medical conditions (E.g. hypotension)
* Frailty due to mental conditions (E.g. dementia)
* Frailty due to physical conditions (E.g. amputation or injury)
* Frailty due to medication(s)

Patients who are able to give informed consent will be included. In addition, any patients who are unable to consent to participation in this study due to a lack of mental capacity but are assessed by the ward matron to benefit from participation in this study will also be included. Where possible, consent will be obtained from close relatives or legal guardians in this case. These patients are a particularly vulnerable group and their interests must therefore be protected. They should be given the same opportunities to participate in ethically designed research projects as those who do not lack capacity but must not be put at unwarranted risk.

Exclusion Criteria:

Patients under 18 years of age Patients who are in an unconscious or comatose state, physically restrained to the bed, or otherwise completely unable to move under their own power and thus not at risk of falling out of their bed

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ward 20 at the Royal Lancaster Infirmary .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-05-03 (Estimated); Primary Completion 2018-08-15 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of falls recorded | 12 months
  The number of falls and fall related incidents in the ward

CONTACTS AND LOCATIONS:
Overall Officials: Kim Wilson, BA (Hons), Principal Investigator — University Hospitals of Morecambe Bay NHS Trust

IPD SHARING:
Plan to Share IPD: No